CLINICAL TRIAL: NCT05136599
Title: Open-label, Phase 1, Dose-escalation Clinical Trial to Establish a Controlled Human Infection Model by Determining the Optimal and Safe Bordetella Pertussis Dose That Induces Mild Symptomatic Infection and Colonization in Healthy Adults
Brief Title: Establishing a Controlled Human Infection Model of Bordetella Pertussis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Centers for Disease Control and Prevention (U.S. Federal Agency); Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CD2001; R34AI148056 (NIH); 75D30120C08608 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2021-11-02; First posted 2021-11-29 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2024-06

CONDITIONS: Pertussis
Keywords: Bordetella pertussis; Pertussis; Whooping cough; Controlled human infection model; Human challenge; Phase 1 clinical trial; Immune response
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Intervention Model Description: The clinical trial will be conducted as two dependent studies. The first study is a dose identification study to determine the HID70-90 endpoint, which is the dose that induces pertussis mild symptomatic/clinical infection among 70%-90% of the volunteers inoculated with that dose. The second study and sub-study are HID70-90 dose confirmation studies to verify and confirm that the infectious endpoint has been reached to establish the pertussis CHIM.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (14):
- Study 1 (Dose-identification study), Cohort 1, Dose #3 (Experimental): Challenge dose of 10^4 cfu B. pertussis in 0.2 mL (0.1 mL per naris)
  Interventions: Biological: Bordetella pertussis D420
- Study 1 (Dose-identification study), Cohort 2, Dose #5 (Experimental): Challenge dose of 10^5 CFU B. pertussis in 0.2 mL (0.1 mL per naris)
  Interventions: Biological: Bordetella pertussis D420
- Study 1 (Dose-identification study), Cohort 3, Dose #6 (Experimental): Challenge dose of 5 x 10^5 CFU B. pertussis in 0.2 mL (0.1 mL per naris)
  Interventions: Biological: Bordetella pertussis D420
- Study 1 (Dose-identification study), Cohort 4, Dose #7 (Experimental): Challenge dose of 10^6 CFU B. pertussis in 0.2 mL (0.1 mL per naris)
  Interventions: Biological: Bordetella pertussis D420
- Study 1 (Dose-identification study), Cohort 5, Dose #8 (Experimental): Challenge dose of 5 x 10^6 CFU B. pertussis in 0.2 mL (0.1 mL per naris)
  Interventions: Biological: Bordetella pertussis D420
- Study 1 (Dose-identification study), Cohort 6, Dose #9 (Experimental): Challenge dose of 10^7 CFU B. pertussis in 0.2 mL (0.1 mL per naris)
  Interventions: Biological: Bordetella pertussis D420
- Study 1 (Dose-identification study), Cohort 7, Dose #9 Repeat (Experimental): Challenge dose of 10^7 CFU B. pertussis in 0.2 mL (0.1 mL per naris)
  Interventions: Biological: Bordetella pertussis D420
- Study 2 (Dose confirmation study), Cohort 8, Dose #9 (Experimental): Challenge dose of 10^7 CFU B. pertussis in 0.2 mL (0.1 mL per naris)
  Interventions: Biological: Bordetella pertussis D420
- Study 2 (Dose confirmation study), Cohort 8, Dose #10 (Experimental): Challenge dose of 5 x 10^7 CFU B. pertussis in 0.2 mL (0.1 mL per naris)
  Interventions: Biological: Bordetella pertussis D420
- Study 2 (Dose confirmation study), Cohort 9, Dose #9 (Experimental): Challenge dose of 10^7 CFU B. pertussis in 0.2 mL (0.1 mL per naris)
  Interventions: Biological: Bordetella pertussis D420
- Study 2 (Dose confirmation study), Cohort 9, Dose #10 (Experimental): Challenge dose of 5 x 10^7 CFU B. pertussis in 0.2 mL (0.1 mL per naris)
  Interventions: Biological: Bordetella pertussis D420
- Study 2 (Dose confirmation study), Cohort 10, Dose #8 (Experimental): Challenge dose of 5 x 10^6 CFU B. pertussis in 0.2 mL (0.1 mL per naris)
  Interventions: Biological: Bordetella pertussis D420
- Study 2 (Dose confirmation study), Cohort 11, Dose #10 (Experimental): Challenge dose of 5 x 10^7 CFU B. pertussis in 0.2 mL (0.1 mL per naris)
  Interventions: Biological: Bordetella pertussis D420
- Sub-Study (Dose confirmation study), Cohort 11, Dose #11 (Experimental): Challenge dose of 10^8 CFU B. pertussis in 0.2 mL (0.1 mL per naris)
  Interventions: Biological: Bordetella pertussis D420

INTERVENTIONS:
Biological: Bordetella pertussis D420 — Intranasal inoculation of Bordetella pertussis D420 in each naris on Day 0 of the study.

SUMMARY:
This study aims to establish a Controlled Human Infection Model of Bordetella pertussis by determining a reproducible and safe infectious bacterial dose (challenge inoculum) that achieves colonization and mild symptomatic infection in healthy adults.

DETAILED DESCRIPTION:
This is a single-center trial to develop a Bordetella pertussis Controlled Human Infection Model (CHIM) using a two-study approach: the first study is a human infectious dose 70%-90% (HID70-90) identification study, and the second an HID70-90 dose confirmation study to verify and confirm that the infectious endpoint has been reached. The infectious endpoint is positive nasopharyngeal culture(s) and/or polymerase chain reaction(s) (PCR(s)) for B. pertussis with concurrent or subsequent development of mild pertussis disease symptoms such as rhinorrhea and cough within the 16-day inpatient period following challenge.

The trial is an open-label, phase 1, dose escalation, self-contained trial; participants will be allocated to challenge dose groups to receive a single intranasal dose of challenge inoculum. All participants will receive a 5-day course of azithromycin eradication therapy either 24-48 hours after they develop symptoms or at the end of the 16-day postchallenge observation period.

The optimal/target inoculum is one that induces mild symptomatic infection and detection of B. pertussis in nasopharyngeal cultures in 70%-90% of participants receiving it, to establish a safe and reproducible pertussis CHIM.

Safety monitoring includes close clinical observation during a 16-21-day inpatient postchallenge period in the Canadian Center for Vaccinology's Challenge Unit, a Data and Safety Monitoring Board, and participant Diary Cards.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, each participant must satisfy ALL of the following criteria:

1. Age 18-40 years, inclusive.
2. Good general health status, as determined by history and physical examination conducted no longer than 30 days prior to the challenge.
3. Participants who, in the opinion of the Investigator, can and will comply with the requirements of the protocol (e.g., complete Diary Cards, return for follow-up visits).
4. Written informed consent obtained from the participant.
5. If female of childbearing potential and heterosexually active, has practiced adequate contraception for 28 days prior to challenge and has a negative pregnancy test on the day before B. pertussis challenge and has agreed to continue adequate contraception until 60 days after inoculation. Adequate contraception is defined as a contraceptive method with a failure rate of <1% per year when used consistently and correctly and, when applicable, in accordance with the product label. Examples include the following:

   * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, or transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, or implantable
   * Intra-uterine device (IUD) with or without hormonal release
   * Vasectomized partner, provided that this is the participant's sole partner and that he has received a medical assessment of the surgical success
   * Credible self-reported history of heterosexual abstinence for at least 28 days prior to challenge
   * Female partner

   A premenopausal woman who has at least one of the following is considered not of childbearing potential:
   * Documented hysterectomy
   * Documented bilateral salpingectomy
   * Documented bilateral oophorectomy
   * Documented and current bilateral tubal ligation or occlusion
6. Currently fully vaccinated against SARS-CoV-2/COVID-19 according to provincial Public Health guidelines.
7. If there is a reported history of SARS-CoV-2/COVID-19 infection, the participant must be asymptomatic for >4 weeks.

Exclusion Criteria:

Participants with ANY of the following criteria at the time of screening will be excluded:

1. Underlying chronic medical condition requiring ongoing follow-up and monitoring by a physician (e.g., diabetes, seizure disorder).
2. Underlying cardiac and/or pulmonary disease including hypertension, angina, prior myocardial infarction, asthma, emphysema, chronic bronchitis, and pulmonary tuberculosis.
3. Moderate or severe symptoms of health anxiety, anxiety, and mood symptoms. Self-reported current diagnosis of a major psychiatric illness, including a schizophrenia spectrum disorder, bipolar disorder, posttraumatic stress disorder, obsessive compulsive disorder, substance use, or eating disorder.
4. QT prolongation on electrocardiogram (EKG).
5. History of everyday smoking/vaping in the last 2 years and/or current smoking/vaping more than once per week.
6. Pregnant (known before or established at the time of screening using a urine-based test) or breastfeeding.
7. Immunocompromised (with HIV/AIDS-positive or receiving immunosuppressive therapy involving steroids) or with any medical condition or medication that leads to a compromised immune system.
8. Positive for hepatitis B or C.
9. Vaccinated against pertussis within previous 5 years and/or >7 cumulative doses from infancy to date of screening.
10. Reported history of laboratory-confirmed pertussis infection.
11. Antibody titer to pertussis toxin >20 EU/mL (2x the lower limit of quantification (LLOQ)).
12. Nasopharyngeal detection of B. pertussis prior to challenge using culture isolation and/or PCR detection, or detection of other respiratory infection.
13. Living with young children (<1 year of age) or with any household member not current in their pertussis immunization up to Day 56 post-challenge. Note: Household members whose vaccination is not current will be offered a pertussis-containing vaccine, as recommended and funded by the Nova Scotia Department of Health and Wellness.
14. Living or working with (any form of close contact) any of the at-risk/vulnerable groups (children <1 year of age, pregnant woman who have not yet received their maternal Tdap vaccine, immunocompromised individuals, anyone not current in their pertussis immunization, or adults >65 years of age who have not received a dose of Tdap vaccine within the past 10 years) up to Day 56 post-challenge.
15. Known allergy to macrolides including azithromycin or erythromycin, history of Clostridium difficile within last 2 months.
16. Any contraindication to receiving azithromycin.
17. Taking any antibiotic currently or within the previous 2 weeks.
18. Currently taking terfenadine, astemizole, theophylline, or cimetidine.
19. Recent (within 6 months) nasal or sinus surgery, recent use of intranasal steroids (4 weeks), or diagnosis with nasal polyps.
20. Receipt of any investigational drug or vaccine (including SARS-CoV-2/COVID-19 vaccine) within 6 months prior to challenge. An investigational vaccine is defined as a vaccine that is still being tested in clinical trials or one that has not yet been authorized for use in Canada for administration by public vaccine programs.
21. Receipt of any authorized vaccines within 2 weeks of being challenged with B. pertussis in this study. (This is to avoid attributing any AEs from these vaccines to the B. pertussis challenge, which would skew the study results.)
22. Current laboratory-confirmed SARS-CoV-2/COVID-19 infection.
23. Previous moderate or severe laboratory-confirmed SARS-CoV-2/COVID-19 infection that required hospitalization.
24. Head trauma (e.g., fracture of the cribriform plate) within 1 year of screening.
25. Any other finding that the Investigator considers will make the participant unsuitable for the study or unable to comply with the study requirements.
26. Symptoms indicative of acute respiratory illness (such as fever, cough, difficulty breathing) identified during the physical examination done on Day -1 (check-in) or Day 0 before a participant is challenged.
27. History of Bell's Palsy and/or facial paralysis.
28. Receipt of facial cosmetic filler in the past 3 months.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with mild symptoms of early pertussis disease postchallenge | Day 0 (challenge day) to Day 16
  Mild, Grade 1, symptoms of pertussis are symptoms that do not interfere with everyday activities. They may include malaise, rhinorrhea, sneezing and/or lacrimation, low-grade fever, or cough.

SECONDARY OUTCOMES:
Number of participants who demonstrate shedding of Bordetella pertussis postchallenge as determined by positive culture and/or PCR test of nasopharyngeal samples | Day 1 to Day 14
  The presence of B. pertussis is detected by positive culture (i.e., presence of any B. pertussis colonies) of nasopharyngeal samples. It is also detected by a positive PCR (polymerase chain reaction) test of nasopharyngeal samples. Both methods are used in this study; a positive result in either culture and/or PCR test demonstrates shedding of B. pertussis.

CONTACTS AND LOCATIONS:
Overall Officials: Scott A. Halperin, MD, Principal Investigator — Dalhousie University
Locations (1):
- Canadian Center for Vaccinology, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Canadian Center for Vaccinology Challenge Unit home page — https://www.challengeunit.ca/
- See also: Canadian Center for Vaccinology home page — http://centerforvaccinology.ca